CLINICAL TRIAL: NCT04661358
Title: A Randomized Clinical Trial Evaluating Fenofibrate for Prevention of Diabetic Retinopathy Worsening
Brief Title: Fenofibrate for Prevention of DR Worsening
Acronym: Protocol AF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH); Juvenile Diabetes Research Foundation (Other); Roche Pharma AG (Industry); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRCR.net Protocol AF; U10EY014231 (NIH)
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Retinopathy
Keywords: Fenofibrate; non-proliferative diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fenofibrate 160-mg (Experimental)
  Interventions: Drug: Fenofibrate
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fenofibrate — Participants begin with a dose of either 160mg or 54mg fenofibrate, based on eGFR value at screening, taken once daily with food. The dose may be adjusted during follow-up based on protocol guidelines.
  Arms: Fenofibrate 160-mg
Other: Placebo — Participants begin with a dose of either 160mg or 54mg placebo, based on eGFR value at screening, taken once daily with food. The dose may be adjusted during follow-up based on protocol guidelines.
  Arms: Placebo

SUMMARY:
This randomized trial will evaluate the effect of fenofibrate compared with placebo for prevention of diabetic retinopathy (DR) worsening through 6 years of follow-up in eyes with mild to moderately severe non-proliferative DR (NPDR) and no CI-DME at baseline.

In addition to evaluating efficacy, this study aims to evaluate the feasibility of a model for ophthalmologists to prescribe or collaborate with a primary care provider such as an internist/endocrinologist to prescribe and monitor the drug safely. If this study demonstrates that fenofibrate is effective for reducing the onset of proliferative diabetic retinopathy (PDR) or and the results are adopted by the community of retina specialists, a new strategy to prevent vision threatening complications of diabetes could be widely adopted. Widespread use of an oral agent effective at reducing worsening of DR would decrease the numbers of patients who undergo more invasive and much more expensive treatment for DR and who are consequently at risk for side effects that adversely affect visual function. This study will also assess the relationship of glycemic variability, as measured by continuous glucose monitoring with DR outcomes. Ancillary studies will characterize functional and structural outcomes in this cohort.

ELIGIBILITY:
Key Inclusion Criteria

* Age ≥18 years and < 80 years.
* Type 1 or type 2 diabetes.
* At least one eye with the following:

  * Mild to moderately severe NPDR (defined by ETDRS DR severity level 35 to 47), confirmed by central Reading Center grading of fundus photographs.
  * Best-corrected E-ETDRS visual acuity letter score of ≥74 (approximate Snellen equivalent 20/32 or better). If best corrected letter score is 74-78, investigator must verify that vision loss is not due to the presence of CI-DME, cataract, or other condition that may affect visual acuity during the course of the study.
* If only one eye is eligible, the non-study eye must have at least microaneurysms only (DR severity level 20)

Key Exclusion Criteria

Eye-level exclusion criteria (the eye is ineligible if any of the following is met):

* Current CI-DME based on clinical exam or OCT central subfield thickness (CST)

  * Zeiss Cirrus: CST ≥290 µm in women or ≥ 305 µm in men
  * Heidelberg Spectralis: CST ≥305 µm in women or ≥320 µm in men
* Any prior treatment for DME or DR, other than focal/grid laser. If the eye has a history of focal/grid laser, it must be at least 12 months prior.
* History of intraocular anti-VEGF or corticosteroid treatment within the prior year for any indication

Participant-level exclusion criterion (the participant is ineligible if the following criterion is met):

• Decreased renal function, defined as requiring dialysis or central laboratory eGFR value < 45 mL/min/1.73 m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Worsening of diabetic retinopathy | 6- years
  Defined as
  * 2 or more step worsening on Early Treatment Diabetic Retinopathy Study (ETDRS) diabetic retinopathy severity on fundus photographs.
  * Development of neovascularization within the 7-modified ETDRS fields on fluorescein angiography.
  * Intraocular procedure undertaken to treat diabetic retinopathy including panretinal photocoagulation, intraocular anti-vascular endothelial growth factor, corticosteroid, or vitrectomy.

SECONDARY OUTCOMES:
Intraocular procedure undertaken to treat diabetic retinopathy or diabetic macular edema including PRP, intraocular anti-VEGF, corticosteroid, focal/grid laser or vitrectomy | 6 years
Development of CI-DME | 6 years
  Defined as, either 1) at least a 10% increase in OCT central subfield thickness from baseline, OCT central subfield thickness greater than sex and machine-specific threshold values (Zeiss Cirrus: CST ≥290 µm in women or ≥ 305 µm in men; Heidelberg Spectralis: CST ≥305 µm in women or ≥320 µm in men), and Investigator determination that thickening cannot be attributed to any cause other than CI-DME, or 2)Intraocular DME treatment including focal/grid laser, intraocular anti-VEGF, intraocular corticosteroid, or vitrectomy
Development of center-involved diabetic macular edema with vision loss | 6 years
  Defined as either 1) an increase in OCT central subfield thickness of 10% or more from baseline, OCT central subfield thickness greater than sex and machine-specific threshold values (Zeiss Cirrus: CST ≥290 µm in women or ≥ 305 µm in men; Heidelberg Spectralis: CST ≥305 µm in women or ≥320 µm in men), investigator determination that thickening cannot be attributed to any cause other than DME, and a decrease in visual acuity from baseline of 10 or more letters at a single visit or 5 to 9 letters at 2 consecutive visits at least 21 days apart with vision loss presumed to be from DME, intraocular DME or 2) treatment including focal/grid laser, anti-VEGF, corticosteroid injection, or vitrectomy
Visual acuity loss from any cause | 6 years
  Defined as a decrease in visual acuity from baseline of 10 or more letters at a single visit or a 5 to 9-letter decrease at 2 consecutive visits at least 21 days apart regardless of whether vision loss is presumed to be from DME or any other cause

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, MD, Study Chair — National Institutes of Health (NIH)
Locations (66):
- United States (66):
  - Kent W. Small, MD, AMC, Glendale, California
  - Salehi Retina Institute Inc., Huntington Beach, California
  - Loma Linda University, Loma Linda, California
  - UCLA Stein Eye Institute, Pasadena, California
  - Regents of the University of California, Davis, DBA University of California, Davis, Sacramento, California
  - The Regents of the University of California, San Francisco, San Francisco, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida- Jacksonville, Jacksonville, Florida
  - Florida Retina Institute, James A. Staman, MD, PA- Jacksonville, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Retina Institute, James A. Staman, MD, PA- Orlando, Orlando, Florida
  - Southeast Eye Institute, P.A. dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Vitreous Consultants, LLP, Sarasota, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - SEASHORE RETINA LLC DBA Retina Specialists of Tampa, Wesley Chapel, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - UIC - Dept of Ophthalmology & Visual Sciences, Chicago, Illinois
  - Illinois Retina Associates SC - Oak Park Site, Oak Park, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - John Kenyon American Eye Institute, LLC, New Albany, Indiana
  - Wolfe Eye Clinic-Cedar Rapids, Hiawatha, Iowa
  - Wolfe Clinic, P.C.- West Des Moines, West Des Moines, Iowa
  - Mid-America Retina Consultants, P.A., Overland Park, Kansas
  - University of Kansas Medical Center Research Institute, Inc., Prairie Village, Kansas
  - Joseph E. Humble and Raymond Haik PTRS DBA Eye Assoc of Northeast Louisiana, West Monroe, Louisiana
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Boston Medical Center Corporation, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Foundation for Vision Research and Retina Specialists of Michigan, P.C., Grand Rapids, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Retina Center, PA DBA Retina Center of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Curators of the University of Missouri, Columbia, Missouri
  - Washington University Ophthalmology, St Louis, Missouri
  - Retina Research Institute, LLC, St Louis, Missouri
  - Retina-Vitreous Surgeons of Central NY, PC, Liverpool, New York
  - MaculaCare, New York, New York
  - Retina Associates of Western NY, P.C., Rochester, New York
  - Pamela Weber, MD/Island Retina, Shirley, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation DBA Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Verum Research LLC, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Retina Consultants, LLC, Salem, Oregon
  - Cascade Medical Research Institute, LLC, Springfield, Oregon
  - Retina-Vitreous Consultants, Inc., Monroeville, Pennsylvania
  - Pittsburg Clinical Trial Consortium, Sewickley, Pennsylvania
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Beaumont, Texas
  - Retina Consultants of Texas, PA, Bellaire, Texas
  - Baylor College of Medicine, Baylor Eye Physicians and Surgeons, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - University of Washington, Seattle, Washington
  - Gunderson Health System, La Crosse, Wisconsin
  - Eye Clinic of Wisconsin, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No